CLINICAL TRIAL: NCT00331682
Title: An Open-Label, Non-Randomized Phase II Study of Alvocidib (Flavopiridol) in Combination With Docetaxel in Refractory, Metastatic Pancreatic Cancer (NCI #6366)
Brief Title: Docetaxel and Flavopiridol in Treating Patients With Refractory Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01471; 05-136; MSKCC-05136; NCI-6366; CDR0000472413; R01CA067819 (NIH)
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2013-11

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — alvocidib; Docetaxel

ARMS (1):
- Treatment (docetaxel and alvocidib) (Experimental): Patients receive docetaxel IV over 30 minutes followed 4-6 hours later by flavopiridol IV over 60 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: alvocidib; Drug: docetaxel

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT

SUMMARY:
Drugs used in chemotherapy, such as docetaxel and flavopiridol, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Flavopiridol may also help docetaxel work better by making tumor cells more sensitive to the drug. This phase II trial is studying how well giving docetaxel followed by flavopiridol works in treating patients with refractory metastatic pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate in patients with refractory, metastatic pancreatic cancer treated with weekly, sequential docetaxel and flavopiridol.

SECONDARY OBJECTIVES:

I. Determine the time to progression and overall survival of patients treated with this regimen.

II. Assess the toxicity of this regimen.

OUTLINE: This is a non-randomized, open-label, prospective study.

Patients receive docetaxel IV over 30 minutes followed 4-6 hours later by flavopiridol IV over 60 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Evidence of metastatic disease
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20mm with conventional techniques or as ≥ 10 mm with spiral CT scan

  * The primary site is not a measurable lesion
* Documented progression with measurable metastatic disease including any 1 of the following criteria:

  * Receiving adjuvant therapy for resected disease
  * Receiving therapy for locally advanced disease
  * Within 3 months of completing adjuvant therapy or therapy for locally advanced disease
  * On 1 prior regimen in the metastatic setting
* No documented brain metastases
* Karnofsky performance status (PS) 80-100% OR ECOG PS 0-1
* WBC ≥ 2,500/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT < 2.5 times ULN
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Alkaline phosphatase ≤ 5 times ULN
* No history of allergic reactions to compounds of similar chemical orbiological composition to flavopiridol
* No known allergy to docetaxel or medications formulated in polysorbate 80 (Tween 80)
* No uncontrolled diabetes
* No uncontrolled intercurrent illness including, but not limited to any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia or myocardial infarction within the past 6 months

    * Rate-controlled atrial fibrillation stable for ≥ 6 months allowed
  * Psychiatric illness or social situations that would limit compliance with study requirements
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No peripheral neuropathy > grade 1
* No immune deficiency
* Atl east 2 weeks since prior chemotherapy (6 weeks for nitrosoureas, carmustine, or mitomycin C) and recovered
* At least 2 weeks since prior targeted therapy (e.g., antiangiogenic therapy [e.g., bevacizumab] or epidermal growth factor receptor [EGFR] tyrosine kinase inhibitor [e.g., erlotinib hydrochloride]) and recovered
* At least 4 weeks since prior radiation therapy
* No prior docetaxel or flavopiridol
* No other concurrent chemotherapy or investigational agents
* No other concurrent anticancer agents or therapies
* No concurrent commonly used vitamins, antioxidants, orherbal preparations or supplements

  * Single-tablet multivitamin allowed
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen O'Reilly, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel and Flavopiridol: Patients receive docetaxel IV over 30 minutes followed 4-6 hours later by flavopiridol IV over 60 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  alvocidib: Given IV
  docetaxel: Given IV
Period: Overall Study
Arm/Group | Docetaxel and Flavopiridol
Started | 10
Completed | 9
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Docetaxel and Flavopiridol: Patients receive docetaxel IV over 30 minutes followed 4-6 hours later by flavopiridol IV over 60 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  flavopiridol: Given IV
  docetaxel: Given IV
Arm/Group | Docetaxel and Flavopiridol
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (21.21320344)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate as Measured by RECIST Criteria
Description: Objective response rate as measured by RECIST criteria
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Docetaxel and Flavopiridol
Number analyzed (Participants) | 9
participants
  Stable Disease | 3
  Progression of Disease | 6

2. Secondary Outcome: Time to Progression
Description: Will be computed using Kaplan-Meier methods.
Time Frame: Between the start of treatment until the criteria for progression are met, assessed up to 2 years
Measure: Median (Full Range); unit: weeks
Arm/Group | Docetaxel and Flavopiridol
Number analyzed (Participants) | 9
weeks | 8 [7 to 14]

3. Secondary Outcome: Overall Survival
Description: Will be computed using Kaplan-Meier methods.
Time Frame: Between the start of treatment until patient death, assessed up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Docetaxel and Flavopiridol
Number analyzed (Participants) | 9
months | 4.2 [2.8 to 6.9]

ADVERSE EVENTS:
Arm/Group | Docetaxel and Flavopiridol
Serious Adverse Events (participants affected / at risk) | 10/10
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel and Flavopiridol (N=10)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Death not associated w/ CTCAE term-Disease Progression NOS (General disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema-visceral (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 4 (4)
Lymphocyte count decreased (Investigations) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (4)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Thrombosis (Vascular disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel and Flavopiridol (N=9)
Alanine aminotransferase increased (Investigations) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (5)
Alkaline phosphatase increased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (9)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 3 (3)
INR increased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 6 (6)
Lymphocyte count decreased (Investigations) | 5 (5)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Platelet count decreased (Investigations) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less